CLINICAL TRIAL: NCT05047328
Title: Early Access Program With Inolimomab in Steroid-refractory Acute Graft Versus Host Disease Grade II-IV in Adults and in Children Over 28 Days of Age
Brief Title: Early Access Program With Inolimomab in Steroid-refractory Acute Graft Versus Host Disease
Status: Available | Type: Expanded Access
Sponsor: ElsaLys Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: ATUC-LKT
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Steroid Resistant Acute Graft Versus Host Disease
MeSH Terms: interventions — inolimomab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: inolimomab — 1 or 2 Induction Phases at 0.3 mg/kg/day for adults or 0.4 mg/kd/day for children over 8 consecutive days If no complete response (CR) occurs after 8 days, a second induction phase is conducted until day 16 (even if CR is obtained before completion of the second induction phase).
  Maintenance Phase: 0.4 mg/kg administered 3 times a week until Day 28 In case of a CR at day 9, the maintenance phase will start after day 9 and will be sustained until day 28.
  In case of a CR, partial response (PR) or mixed response (MR) at day 17, the maintenance phase will start after day 17 and will be sustained until day 28.
  Total duration of treatment is 28 ±2 days.
  Other Names: Leukotac

SUMMARY:
Leukotac (inolimomab) is not approved yet for marketing in any region. In the absence of medical options and based on the safety and efficacy data obtained during the clinical development program (in a phase III (INO-107) and in a Long Term Follow Up study), the French National Agency for the Medicines and Health Products Safety (ANSM) granted a Temporary Authorisation for Use (ATU) so-called cohort ATU (cATU) for LEUKOTAC® (inolimomab) and approved the temporary use protocol .

This early access program has been granted to Leukotac (inolimomab) in adults and in children over 28 days of age, for treatment of acute cortico-resistant or cortico-dependent grades II-IV acute graft versus host disease (GvHD) according to the Glucksberg classification after allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Despite improvements in allogeneic hematopoietic stem cell transplantation (allo-HSCT) settings, graft-versus-host disease (GvHD) remains a significant issue after transplantation and a major cause of non-relapse mortality. Acute GvHD (aGvHD) still develops in about 30% to 80% of patients, for which high dose corticosteroids can be initiated in those with grade ≥II. However, up to 50% of patients fail to obtain a satisfactory response with steroid treatment alone. Treatment of steroid-resistant (SR) aGvHD remains an unmet clinical need.

Inolimomab is an IgG1 mouse monoclonal antibody which specifically binds to the alpha chain of the human interleukin-2 receptor (CD25, IL-2R), a receptor expressed on the surface of the T cells in response in to antigenic stimulation.

Inolimomab efficacy in the treatment of corticosteroid-resistant graft-versus-host disease after allogenic hematopoietic stem cell transplant was assessed in a multicenter phase 3 randomized double-blind controlled study (INO-0107) versus Thymoglobulin® (anti-thymocyte globulin (ATG )).

Long term survival data were collected in the 43 surviving patients at the end of the phase 3 study INO-0107 (23 inolimomab; 20 ATG) and up to 104 months after discontinuation of treatment (median follow-up: 58.4 months). These long term follow-up data showed a statistically significant difference for survival with relative risk of death reduced by 43% in the inolimomab group (p=0.030). These data confirm the 1-year observations of the phase 3 study INO-0107 with a clear clinical benefit on survival statistically greater in patients receiving inolimomab.

Leukotac (inolimomab) is not approved yet for marketing in any region. This early access program has been granted to Leukotac (inolimomab) in adults and in children over 28 days of age, for treatment of acute cortico-resistant or cortico-dependent grades II-IV acute graft versus host disease (GvHD) according to the Glucksberg classification after allogeneic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 28 days
* Grade II-IV acute graft versus host disease according to Glucksberg classification after allogeneic hematopoietic stem cell transplantation
* Patients resistant or dependent to corticosteroid (CS)

Exclusion Criteria:

* Pregnancy
* Breastfeeding

Min Age: 28 Days | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- ElsaLys Biotech, Lyon, France